CLINICAL TRIAL: NCT06319573
Title: Evaluation of in Vitro Fertilisation Patients' Experience With a Personalized Prognostic Counseling Strategy and Its Impact on Treatment Utilization and Discontinuation
Brief Title: The Impact of Personalized Prognostic Counseling on IVF Patient's Experience and Treatment Utilization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ginefiv (Other)
Collaborators: Univfy Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2305-UNIVF-070-DC
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Infertility
Keywords: Infertile Women Undergoing IVF or ICSI; Fertility Issues; Machine Learning; Counseling
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Counseling (Active Comparator): Patients in this group will be counseled as per standard care during their second consultation. They will be asked to complete an anonymous online validated questionnaire (see below) to assess their responses to the anonymous online questionnaire after consultation.
  Interventions: Other: Standard Counseling
- Counseling Supported by Univfy® Report (Experimental): Patients in this group will be counseled with the Univfy® PreIVF report during their second consultation. They will also be asked to fill out the same anonymous online questionnaire.
  Interventions: Other: Counseling Supported by Univfy® Report

INTERVENTIONS:
Other: Counseling Supported by Univfy® Report — The intervention consists of patients being counseled with the Univfy® PreIVF report during their second consultation. They will also be asked to fill in the same anonymous online questionnaire.
  Arms: Counseling Supported by Univfy® Report
Other: Standard Counseling — Patients in this group will be counseled as per standard care during their second consultation. They will be asked to complete an anonymous online validated questionnaire (see below) to assess their responses to the anonymous online questionnaire after consultation.
  Arms: Standard Counseling

SUMMARY:
This study will be conducted in two phases. In the first phase, research subjects will be assigned to receive standard counseling. In the second phase, research subjects will receive Univfy counseling.

DETAILED DESCRIPTION:
Study period: 6 months plus 12 months follow-up. Participating centers: Ginefiv Madrid and Barcelona Inclusion / Exclusion criteria: See the Section on Inclusion and Exclusion Criteria.

In the first three months of the study, the participants (consenting patients) will be counseled as per standard care during their consultations ("Phase 1: Standard Counseling"). They will be asked to complete an anonymous online questionnaire to assess their experience after the consultation.

In the following 3 months of the study ("Phase 2: Univfy Report"), the participants (different from participants recruited in Phase 1) will instead be counseled with the Univfy PreIVF report during their initial consultation or subsequent consultations (as soon as a Univfy PreIVF report can be generated). They will be asked to complete an anonymous online questionnaire to assess their experience after the consultation.

During the following 12 months ("Phase 3: Outcomes Data Collection Period"), we will measure 1) patient experience based on patients' responses to the anonymous online questionnaire 2) IVF and intrauterine insemination (IUI) treatment utilization rates within 6 and 12 months, 3) patient retention rates after the first failed treatment attempt, 4) IUI-live birth rates and the cumulative live birth delivery rate (CLBdR, defined according to ICMART). The above metrics will be compared between participants who received conventional counseling versus those who received the Univfy report.

Outcomes:

* IUI and IVF treatment utilization (conversion) rates in the two groups
* Responses to the anonymous online questionnaire in the two groups
* Retention rate in the two groups
* Time to pregnancy

Sub-analyses will be conducted in different patient populations (e.g., poor responders, severe male factor, the indication to PGT-A) and according to each IVF center and clinician. Here are categories defined a priori that will be used in sub-group analysis: prognostic tier, with each tier defined by the PreIVF model-predicted probability of live birth (this is the most objective way to define a sub-group)

* Age
* AMH levels
* BMI values
* clinical diagnoses such as male factor, poor ovarian response/reserve, tuba! factor, uterine factor, endometriosis, etc.

Interim Analysis:

Interim analyses will be conducted at Month#9, Month#12, Month#15, and Month#18 to allow identification of positive results should they occur prior to the completion of Phase 2. Physicians will be blinded to the results of the analysis.

Sample size analysis:

Estimating a 15%-increase in the treatment conversion rate (from 50 to 65%) with 80% power and 5% alpha error probability, we will need at least 183 patients per group (366 in total).

Estimating a 20%-decrease in the treatment discontinuation between first, and second attempts (from 70 to 50%) with 80% power and 5% alpha error probability, we will need at least 102 patients who failed a first attempt per group (204 in total).

Univfy® products and services are protected by US Patent Number 9,458,495B2, foreign counterparts and other issued and pending patents.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-43 in age and their healthcare providers have determined that IVF treatment using the patients' own eggs is indicated.

Exclusion Criteria:specific to this study only (these are not contraindications to using the Univfy® PreIVF Report):

* Same sex couples
* Patients undergoing DuoStim and/or PGT-M/-SR
* Patients considering egg freezing rather than IVF
* Patients considering the use of donor eggs or gestational carrier

Patients with contraindications to receiving the Univfy® PreIVF Report For Patients Under 40 Using Their Own Eggs. Those contraindications are:

* Patients who are perimenopausal or menopausal
* Patients who have very poor IVF results in the past, including:
* extremely poor oocyte/embryo quality, no embryos to transfer,
* no euploid embryos on PGT-A, no blastocysts in extended culture

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 366 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Treatment utilization (conversion) rate in the two groups | A full 12 months of follow up starting at the end of Phase 2. An interim analysis using data up to the 6 months following the end of Phase 2 will be performed .
  The treatment conversion rate refers to the proportion of patients who initiate IVF treatment after undergoing the initial consultation and counseling. This outcome will be compared between the two groups.
Patient experience responses | A full 12 months of follow up starting at the end of Phase 2. An interim analysis using data up to the 6 months following the end of Phase 2 will be performed
  Research satisfaction topics related to counseling about IVF treatment and IVF treatment success probability on a scale of 1-5:
  Consultation met expectations Satisfied with explanation of consent Felt listened to by your physician Satisfied with physician's explanation of treatment needed Satisfied with physician's explanation of medications needed and possible side effects Satisfied with clarity of physician's explanation of probability of IVF success Satisfied with material given to explain probability of IVF success Your physician's clarity and honesty about your probability of IVF success Do you think receiving information about your chances of treatment failure will help you to cope with the whole treatment.
Validation of Univfy prediction upon CLBdR | A full 12 months of follow up starting at the end of Phase 2. An interim analysis using data (e.g. positive serum HCG, fetal sac on ultrasound, fetal heart on ultrasound) up to the 6 months following the end of Phase 2 will be performed . Study follow up
  This outcome assesses the accuracy of the Univfy model's predictions regarding cumulative live birth delivery rate (CLBdR). It compares the predicted CLBdR for each patient group with their actual CLBdR after completing the treatment cycle.
Retention Rate | A full 12 months of follow up starting at the end of Phase 2. An interim analysis using data up to the 6 months following the end of Phase 2 will be performed
  This outcome measures the proportion of patients who continue with IVF treatment attempts after facing an unsuccessful first cycle.
Time to Pregnancy | A full 12 months of follow up starting at the end of Phase 2. An interim analysis using data up to the 6 months following the end of Phase 2 will be performed .
  This outcome tracks the duration it takes for a patient to achieve pregnancy after the initial and second consultation.

SECONDARY OUTCOMES:
Self-reported satisfaction related to psychological support and cost of treatment | A full 12 months of follow up starting at the end of Phase 2. An interim analysis using data up to the 6 months following the end of Phase 2 will be performed .
  Research satisfaction topics based on patient's self-reported satisfaction related to psychological support and cost of treatment on a scale of 1-5:
  Satisfied with the level of attention given to your emotional needs Satisfied with the explanation given on the cost of treatment Satisfied with the time of the first visit Satisfied with the way your physician proposed psychological support Do you believe that psychological support is important after being diagnosed with infertility

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Ginefiv S.L, Barcelona
  - Ginefiv S.L, Madrid

IPD SHARING:
Plan to Share IPD: No